CLINICAL TRIAL: NCT02903030
Title: Probiotics for Quality of Life in Autism Spectrum Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Autism Treatment Network (Network); Autism Speaks (Other)
Responsible Party: Principal Investigator, L. Eugene Arnold, Professor Emeritus of Psychiatry, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016H0174
Record Dates: First submitted 2016-06-14; First posted 2016-09-16 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Autism Spectrum Disorders; Anxiety
Keywords: Gastrointestinal Microbiome
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders | interventions — Maltose; Silicon Dioxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Visbiome, Then Placebo (Experimental): The probiotic mix (VISBIOME) will be mainly Bifidobacteria and Lactobacilli, in view of the previously reported encouraging clinical studies and safety data.
  Interventions: Drug: Visbiome Extra Strength
- Placebo, Then Visbiome (Placebo Comparator): Placebo matched to probiotic.
  Interventions: Drug: Maltose (placebo)

INTERVENTIONS:
Drug: Maltose (placebo) — Maltose with a trace amount of silicon dioxide
  Other Names: Maltose with silicon dioxide
  Arms: Placebo, Then Visbiome
Drug: Visbiome Extra Strength — It is a mix of 8 strains of beneficial bacteria that should improve gut flora, improving GI function and hopefully anxiety
  Arms: Visbiome, Then Placebo

SUMMARY:
A randomized pilot trial of a probiotic for quality of life in autism spectrum disorder (ASD), targeting gastrointestinal (GI) symptoms.

DETAILED DESCRIPTION:
The physical and mental/emotional health of people with autism spectrum disorder (ASD) are closely connected. The emerging data on immune abnormalities and gut microbiome differences, and interactions of the genome with these suggest a possible etiological link between physical and mental dysfunction, especially the gastrointestinal (GI) dysfunction and severe anxiety that many individuals with ASD manifest. The investigators have preliminary clinical evidence that children with ASD & GI symptoms differ in microbiome composition and function from neurotypical children with GI symptoms. The investigators hypothesize that altered host-microbial signals, which include altered fecal neurotransmitter gamma-aminobutyric acid (GABA) levels contribute towards anxiety and sensory over-responsivity in ASD. Our preliminary findings also show that probiotic Visbiome Extra Strength, improves GI and pain symptoms, correlating with altered gut microbiome composition and related metabolites (the macrobiome). The proposed crossover trial will explore the possibilities of this new appreciation of the microbiome-mental/physical function connection for ASD, GI dysfunction, and anxiety. If altering the gut microbiome results in better GI and emotional function, it could improve the quality of life for children with ASD and their parents. A pilot trial with 12 children with ASD will test feasibility for a proposed three-site crossover randomized clinical trial (RCT) of probiotics (beneficial bacteria including Lactobacilli & Bifidobacteria) in 60 children 3-12 years old with ASD, GI dysfunction, & anxiety. In a balanced crossover children will be randomized 1;1 to Visbiome or placebo first, 8 weeks per condition with 3 weeks washout between. The investigators have access to significant fecal microbiome and metabolome data from NIH-funded Human Microbiome Projects (HMP) on similar-age healthy and irritable-bowel children, with and without ASD. These will help leverage our understanding of macrobiome changes that correlate with functional improvement of GI and abdominal pain symptoms. Pilot study efficiency will also benefit from those HMPs having already collected and analyzed baseline stools for some children with ASD, thus saving significant costs for baseline stool analyses for the pilot.

ELIGIBILITY:
Inclusion Criteria:

1. have DSM-5 ASD on clinical evaluation by a doctoral-level diagnostician, confirmed by Autism Diagnostic Interview-Revised or Autism Diagnostic Observation Schedule;
2. be between 3 and 12 years old;
3. have >2 mo. abdominal pain, constipation, diarrhea, and/or vomiting, with an item-mean score >2 on at least one scale of the GI module of the PedsQL scale;
4. have clinical anxiety symptoms with an item mean of >1.0 (0-3 scale) on the new Autism Anxiety Scale.

Participants will be recruited from minority, poor, inner city, or rural populations.

Exclusion Criteria:

1. Antibiotics in 2 months prior to enrolling;
2. Prior bowel surgery;
3. Chronic serious medical condition (e.g., diabetes);
4. Weight or height < 3rd %ile for age;
5. Chronic anti-inflammatory use within 2 months prior to enrolling;
6. History of inflammatory bowel disease, Celiac disease, or eosinophilic disorders (e.g., eosinophilic esophagitis);
7. Already taking probiotics within the previous 6 months.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Arnold, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 participants were screened and randomized to be in the study at the OSU Wexner Medical Center, Nisonger Center in 2016.
Pre-assignment Details: 13 patients were randomized to order, but 3 dropped out because of distance and transportation without providing any follow-up data, leaving 10 who progressed through to study completion. (77% retention rate)
Groups:
- Visbiome, Then Placebo: Children aged 3-12 years with ASD, GI symptoms, and anxiety were randomly assigned 1:1 to probiotic Visbiome for 8 weeks, followed by a 3-week washout and an 8 week crossover treatment (19 weeks total).
  The probiotic mix (VISBIOME) will be mainly Bifidobacteria and Lactobacilli, in view of the previously reported encouraging clinical studies and safety data.
  Visbiome Extra Strength: It is a mix of 8 strains of beneficial bacteria that should improve gut flora, improving GI function and hopefully anxiety
- Placebo, Then Visbiome: Children aged 3-12 years with ASD, GI symptoms, and anxiety were randomly assigned 1:1 to placebo for 8 weeks, followed by a 3-week washout and an 8 week crossover treatment (19 weeks total).
  Placebo matched to probiotic.
  Maltose (placebo): Maltose with a trace amount of silicon dioxide
Period: First Intervention (8 Weeks)
Arm/Group | Visbiome, Then Placebo | Placebo, Then Visbiome
Started | 8 | 5
Received Intervention | 6 | 4
Completed | 6 | 4
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: Washout (3 Weeks)
Arm/Group | Visbiome, Then Placebo | Placebo, Then Visbiome
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Visbiome, Then Placebo | Placebo, Then Visbiome
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- Visbiome, Then Placebo: Participants were randomly assigned 1:1 to Visbiome probiotic for 8 weeks, followed by a 3-week washout and an 8 week crossover treatment. (19 weeks total) Starting dose: the first 4 weeks, was a half packet twice daily mixed with food. At 4 week and 15-week visit, there was an option to increase to a full packet twice daily if no effect was noted.
  The probiotic mix (VISBIOME) will be mainly Bifidobacteria and Lactobacilli, in view of the previously reported encouraging clinical studies and safety data.
  Visbiome Extra Strength: It is a mix of 8 strains of beneficial bacteria that should improve gut flora, improving GI function and hopefully anxiety
- Placebo, the Visbiome: Particiapants were randomly assigned 1:1 to placebo for 8 weeks, followed by a 3-week washout and an 8 week crossover treatment. (19 weeks total) Starting dose: the first 4 weeks of the probiotic treatment was a half packet twice daily mixed with food. At 4 week and 15-week visit, there was an option to increase to a full packet twice daily if no effect was noted.
  Placebo matched to probiotic.
  Maltose (placebo): Maltose with a trace amount of silicon dioxide
- Total: Total of all reporting groups
Arm/Group | Visbiome, Then Placebo | Placebo, the Visbiome | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 10
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 2 | 1 | 3
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10
Gastrointestinal Module of the Pediatric Quality of Life Inventory (PedsQL) [Mean (Standard Deviation); unit: units on a scale] — A 74-item survey with 14 scales. Report forms for specific age ranges assess the parent's perception of the child's GI function and/or symptoms during the last month on a 5-point scale from 0 (never a problem) to 4 (almost always a problem). Items are reverse-scored and transformed to a 0-100 scale so lower scores reflect worse GI dysfunction. Response choices are in Likert-scale format ranging from 0 to 4 (0=Never, 1=Almost Never, 2=Sometimes, 3=Often, 4=Almost Always).
  units on a scale | 66.73 (20.193) | 59.60 (17.214) | 63.17 (18.76)
Parent-Rated Anxiety Scale for ASD (PRAS-ASD) [Mean (Standard Deviation); unit: units on a scale] — A 25-item single-factor scale measure of emotional stability/anxiety summed to get a score. Higher scores are worse for PRAS-ASD subscale. Scores range from 0-75.
  units on a scale | 40.00 (15.582) | 41.25 (10.012) | 40.63 (18.52)
Aberrant Behavior Checklist (ABC) [Mean (Standard Deviation); unit: units on a scale] — The ABC is a 58-item parent rating on a 0-3 scale with five subscales:
  1. . Irritability (includes agitation, aggression, and self-injury, 15 items) with range of scores from 0-45
  2. . Social Withdrawal (16 items) with range of scores from 0-48
  3. . Stereotypies (7 items) with range of scores from 0-21
  4. . Hyperactivity (16 items) with range of scores from 0-48
  5. . Inappropriate Speech (4 items) with range of scores from 0-12.
  Higher scores are worse for the ABC subscale.
  units on a scale
    (1) irritability | 18.50 (12.661) | 25.00 (10.801) | 21.75 (16.64)
    (2) lethargy | 18.83 (12.336) | 21.25 (13.598) | 20.04 (18.35)
    (3) stereotypy | 9.33 (4.803) | 10.00 (8.287) | 9.67 (9.57)
    (4) hyperactivity | 22.67 (11.639) | 35.00 (10.132) | 28.83 (15.43)
    inappropriate speech | 5.33 (3.327) | 8.25 (4.500) | 6.79 (5.60)
Social Responsiveness Scale (SRS) [Mean (Standard Deviation); unit: units on a scale] — This 65-item rating scale measures the severity of autism spectrum symptoms as they occur in natural social settings. The SRS provides a clear picture of a child's social impairments, assessing social awareness, social information processing, capacity for reciprocal social communication, social anxiety/avoidance, and autistic preoccupations and traits. It is appropriate for use with children from 4 to 18 years of age and will detect changes in core ASD symptoms. A higher score in this scale represents worse symptoms with raw scores summed and generated t-scores ranging from 0-110.
  units on a scale | 82.17 (7.859) | 87.00 (4.761) | 84.585 (9.189)
Abbreviated Children's Sleep Habits Questionnaire (CSHQ) [Mean (Standard Deviation); unit: units on a scale] — It includes 33 items rated retrospectively over the previous week by parents yielding a total score and eight subscales. Eight subscales include: (1) bedtime resistance (2) sleep onset latency, (3) sleep duration, (4) anxiety around sleep, (5) night awakenings, (6) sleep disordered breathing, (7) parasomnias and (8) morning waking/daytime sleepiness.Total score (summed) range of 0-99. A higher score is a better outcome for this measure.
  units on a scale | 43.50 (8.02) | 59.75 (13.00) | 51.63 (15.27)
Parenting Stress Index Short Form (PSI) [Mean (Standard Deviation); unit: units on a scale] — The PSI is used to evaluate the degree of stress in the parent-child relationship. The Short Form has 36 items from the full length PSI, rated on a 5-point scale from 1 = strongly disagree, to 5 = strongly agree. It is completed in 10-15 minutes. The PSI may be used for parents of children up to 12 years. It yields a Total Score and three domain scores. This will detect effect on parental stress and QOL. Higher scores are worse for the PSI with sums ranging from 0-180.
  units on a scale | 108.17 (20.731) | 129.50 (17.767) | 118.84 (27.303)

OUTCOME MEASURES:

1. Primary Outcome: Change in Gastrointestinal (GI) Module of the Pediatric Quality of Life Inventory (PedsQL) at From Baseline at Week 8
Description: A 74-item survey with 14 scales. Report forms for specific age ranges assess the parent's perception of the child's GI function and/or symptoms during the last month on a 5-point scale from 0 (never a problem) to 4 (almost always a problem). Items are reverse-scored and transformed to a 0-100 scale so lower scores reflect worse GI dysfunction. Response choices are in Likert-scale format ranging from 0 to 4 (0=Never, 1=Almost Never, 2=Sometimes, 3=Often, 4=Almost Always).
Time Frame: Baseline and Week 8 of Both the First and Second Intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Visbiome: Randomly assigned 1:1 probiotic for 8 weeks, followed by a 3-week washout and an 8 week crossover treatment. (19 weeks total) Starting dose, the first 4 weeks, was a half packet twice daily mixed with food. At 4 week and 15-week visit, there was an option to increase to a full packet twice daily if no effect was noted.
  The probiotic mix (VISBIOME) will be mainly Bifidobacteria and Lactobacilli, in view of the previously reported encouraging clinical studies and safety data.
  Visbiome Extra Strength: It is a mix of 8 strains of beneficial bacteria that should improve gut flora, improving GI function and hopefully anxiety
- Placebo: Randomly assigned 1:1 placebo for 8 weeks, followed by a 3-week washout and an 8 week crossover treatment. (19 weeks total) Starting dose, the first 4 weeks, was a half packet twice daily mixed with food. At 4 week and 15-week visit, there was an option to increase to a full packet twice daily if no effect was noted.
  Placebo matched to probiotic.
  Maltose (placebo): Maltose with a trace amount of silicon dioxide
Arm/Group | Visbiome | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale | 17.97 (14.105) | 7.98 (11.247)

2. Secondary Outcome: Change in Target Symptom Rating From Baseline at Week 8
Description: Parents are asked to name the 2 problems of most concern to them at baseline; a clinician helps the parent quantify and describe the problem (frequency, duration, severity, interference with daily life) at baseline. At subsequent visits the clinician reminds the parent of the previous description and helps them again quantify/describe the current state. A panel of blind clinicians reviews the descriptions and rates each on a 9-point scale relative to baseline, from remission (0) to disastrously worse (9), with 5=no change. These ratings are averaged, capturing the issues of most concern to parents across families. For purposes of this study, one of the 2 problems will be required to pertain to GI function, and will be analyzed separately as well as being averaged into the overall symptom rating.
Time Frame: Baseline and Week 8 of Both the First and Second Intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Visbiome: The probiotic mix (VISBIOME) will be mainly Bifidobacteria and Lactobacilli, in view of the previously reported encouraging clinical studies and safety data.
  Visbiome Extra Strength: It is a mix of 8 strains of beneficial bacteria that should improve gut flora, improving GI function and hopefully anxiety
- Placebo: Placebo matched to probiotic.
  Maltose (placebo): Maltose with a trace amount of silicon dioxide
Arm/Group | Visbiome | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale | -2.10 (1.647) | -0.60 (1.370)

3. Secondary Outcome: Change in Parent Anxiety Checklist--ASD From Baseline at Week 8
Description: A 25-item single-factor scale measure of emotional stability/anxiety. Higher scores are worse for PRAS-ASD subscale, hence a negative estimate means more improvement with the probiotics compared to control. Scores range from 0-75.
Time Frame: Baseline and Week 8 of Both the First and Second Intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Visbiome | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale | -6.20 (10.830) | -4.10 (11.259)

4. Secondary Outcome: Change in The Aberrant Behavior Checklist (ABC) From Baseline at Week 8
Description: The ABC is a 58-item parent rating on a 0-3 scale with five subscales:
  * Irritability (includes agitation, aggression, and self-injury, 15 items) with range of scores from 0-45
  * Social Withdrawal (16 items) with range of scores from 0-48
  * Stereotypies (7 items) with range of scores from 0-21
  * Hyperactivity (16 items) with range of scores from 0-48
  * Inappropriate Speech (4 items) with range of scores from 0-12.
  Higher scores are worse for the ABC subscale, hence a negative estimate means more improvement with the probiotics compared to control.
Time Frame: Baseline and Week 8 of Both the First and Second Intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Visbiome | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale
  ABC (1) Irritability | -1.80 (5.245) | -3.50 (5.622)
  ABC (2) Lethargy | -2.60 (8.140) | -2.50 (4.327)
  ABC (3) Stereotypy | -1.20 (4.367) | -1.80 (3.521)
  ABC (4) Hyperactivity | -2.10 (6.385) | -5.40 (6.851)
  ABC (5) Inappropriate Speech | -0.40 (2.011) | -0.10 (1.370)

5. Secondary Outcome: Change in Social Responsiveness Scale (SRS) From Baseline at Week 8
Description: This 65-item rating scale measures the severity of autism spectrum symptoms as they occur in natural social settings. The SRS provides a clear picture of a child's social impairments, assessing social awareness, social information processing, capacity for reciprocal social communication, social anxiety/avoidance, and autistic preoccupations and traits. It is appropriate for use with children from 4 to 18 years of age and will detect changes in core ASD symptoms. A higher score in this scale represents worse symptoms with raw scores summed and generated t-scores ranging from 0-110.
Time Frame: Baseline and Week 8 of Both the First and Second Intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Visbiome | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale | -4.70 (6.255) | -1.70 (5.187)

6. Secondary Outcome: Children's Sleep Habits Questionnaire (CSHQ) at Week 8
Description: It includes 33 items rated retrospectively over the previous week by parents yielding a total score and eight subscales. Eight subscales include: (1) bedtime resistance (2) sleep onset latency, (3) sleep duration, (4) anxiety around sleep, (5) night awakenings, (6) sleep disordered breathing, (7) parasomnias and (8) morning waking/daytime sleepiness.Total score (summed) range of 0-99. A higher score is a better outcome for this measure.
Time Frame: Week 8 of Both the First and Second Intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Visbiome | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale | 42.80 (7.510) | 43.44 (7.502)

7. Secondary Outcome: Change in The Parenting Stress Index Short Form (PSI)
Description: The PSI is used to evaluate the degree of stress in the parent-child relationship. The Short Form has 36 items from the full length PSI, rated on a 5-point scale from 1 = strongly disagree, to 5 = strongly agree. It is completed in 10-15 minutes. The PSI may be used for parents of children up to 12 years. It yields a Total Score and three domain scores. This will detect effect on parental stress and QOL. Higher scores (ranging from 0-180) are worse for PSI, hence a negative estimate means more improvement with the probiotics compared to control.
Time Frame: Baseline and Week 8 of Both the First and Second Intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Visbiome | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale | -9.60 (16.675) | -1.70 (5.187)

ADVERSE EVENTS:
Time Frame: After Baseline: 4 weeks, 8 weeks, 15 weeks, 19 weeks
Description: Collected AE data from all participants of the study.
Groups:
- Visbiome: Randomly assigned 1:1 probiotic for 8 weeks, followed by a 3-week washout and an 8 week crossover treatment. (19 weeks total) Starting dose, the first 4 weeks, was a half packet twice daily mixed with food. At 4 week and 15-week visit, there was an option to increase to a full packet twice daily if no effect was noted.
  The probiotic mix (VISBIOME) will be mainly Bifidobacteria and Lactobacilli, in view of the previously reported encouraging clinical studies and safety data.
  Visbiome Extra Strength: A mix of 8 strains of beneficial bacteria that should improve gut flora, improving GI function and hopefully anxiety
Arm/Group | Visbiome | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visbiome (N=10) | Placebo (N=10)
Gastrointestinal Disorders (Gastrointestinal disorders) | 6 (7) | 4 (9) — Abdominal distension (S:1, P:1)** Abdominal pain (S:1 P:2) Diarrhoea (S:0 P:2) Flatulence (S:3 P:2) Nausea (S:1 P:2) Vomiting (S:1 P:0) ** S= Supplement/Probiotic P = Placebo number is events reported

LIMITATIONS AND CAVEATS:
Small sample. Crossover did not accurately anticipate the duration of carryover Crossover not the best design for this treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT02903030/Prot_SAP_000.pdf